CLINICAL TRIAL: NCT02112318
Title: Study of ECG-derived Atrial Fibrillatory Rate for Prediction of the Outcome of Cardioversion of Short Duration Atrial Fibrillation
Brief Title: CArdioversion of Short Duration Atrial Fibrillation
Acronym: CASAF
Status: Terminated | Type: Observational
Why Stopped: Opposite trend after interim analysis
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: CASAF20090610
Record Dates: First submitted 2014-03-26; First posted 2014-04-11 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation; Electrocardiography; Electrical Remodeling
MeSH Terms: conditions — Atrial Fibrillation; Atrial Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The study is aimed at testing the hypothesis whether atrial fibrillary rate (AFR), as a measure of atrial electrical remodeling assessed from surface ECG, is predictive of sinus rhythm maintenance after electrical cardioversion.

Earlier studies performed in a retrospective fashion suggested that high AFR exceeding 350-360 fibrillations per minute is an independent predictor of AF relapse after cardioversion, particularly in patients with duration of AF episode not exceeding 30 days, however this hypothesis has not been tested in a prospective study.

CASAF is an observational study that will enroll patients with short duration (< 30 days) AF admitted for electrical cardioversion. Admission ECG will be extracted in a digital format and processed off-line for estimation of AFR. AF relapse will be assessed during 6-weeks long follow-up period during which ECG control will be scheduled at week 1 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent AF verified by at least one ECG recording prior to the index admission
* Known onset of symptoms within 30 days from index admission.
* Sinus rhythm ECG within 30 days prior to the index admission If onset of symptoms is unknown.
* If duration of the present AF episode >48 hours then thromboembolic risk should be minimized by either verifying that the patient is adequately anticoagulated according to the hospital routine or TEE performed to verify the lack of contraindications for electrical cardioversion.
* Echocardiography at any time since first onset of AF to verify the lack of significant valvular disease.
* Age older than 18 years.

Exclusion Criteria:

* AF due to reversible cause or significant valvular heart disease
* Treatment with class I or III antiarrhythmic drugs within five half-lives of their elimination period. No amiodarone treatment within six months before admission
* Prior ablation of AF
* Unability to verify onset of symptoms within 30 days prior to the index admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recent onset persistent atrial fibrillation admitted for cardioversion
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Documentation of atrial fibrillation by ECG during follow up period after cardioversion | 6 weeks
  Primary outcome measure in the CASAF study is the number of patients who had relapse of atrial fibrillation during follow up. Primary analysis will be based on assessment the value of the ECG-derived atrial fibrillary rate < vs >= 350 f.p.m. for prediction of atrial fibrillation relapse during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Pyotr G Platonov, MD, PhD, Principal Investigator — Lund University
Locations (3):
- l'Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada
- Sweden (2):
  - Kristianstad General Hospital, Kristianstad
  - Skane University Hospital, Lund

REFERENCES:
- [Background] Holmqvist F, Stridh M, Waktare JE, Sornmo L, Olsson SB, Meurling CJ. Atrial fibrillatory rate and sinus rhythm maintenance in patients undergoing cardioversion of persistent atrial fibrillation. Eur Heart J. 2006 Sep;27(18):2201-7. doi: 10.1093/eurheartj/ehl098. Epub 2006 Sep 6. PMID 16956916
- [Background] Choudhary MB, Holmqvist F, Carlson J, Nilsson HJ, Roijer A, Platonov PG. Low atrial fibrillatory rate is associated with spontaneous conversion of recent-onset atrial fibrillation. Europace. 2013 Oct;15(10):1445-52. doi: 10.1093/europace/eut057. Epub 2013 Mar 20. PMID 23515337
- [Result] Holmqvist F, Seifert MB, Fagerstrom VL, Nault I, Ostenson S, Carlson J, Ekelund U, Platonov PG. Study of ECG-derived atrial fibrillatory rate for prediction of the outcome of cardioversion of short duration atrial fibrillation (CASAF). J Electrocardiol. 2023 Nov-Dec;81:20-22. doi: 10.1016/j.jelectrocard.2023.07.003. Epub 2023 Jul 14. PMID 37480800